CLINICAL TRIAL: NCT01397383
Title: The Effect of Serum Vitamin D Level and the Short Term Functional Outcomes After Total Hip Arthroplasty
Brief Title: Vitamin D and Functional Outcomes After Total Hip Arthroplasty (THA)
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 10014
Record Dates: First submitted 2011-07-15; First posted 2011-07-19 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Vitamin D deficiency: Patients with low serum vitamin D (25-hydroxy vitamin D < 32 ng/ml)
- Control group: Patients with normal serum vitamin D level (serum 25-hydroxy vitamin D > 32 ng/ml)

SUMMARY:
The investigators would like to evaluate the effect of serum 25-hydroxy vitamin D level on post-operative short-term functional outcomes after total hip arthroplasty (THA).

Hypothesis: Patients with low serum vitamin D level will have less within-patient improvement in pre- to 6 week, 1 year, 2 year and 5 year post THA WOMAC scores, SF-36 scores, and performance-based tests(get up and go test and 2 minute walking test) compared to patients who do not have a low vitamin D levels.

Also, Patients with low serum vitamin D level will have a higher rate of postoperative thigh pain or periprosthetic fracture.

DETAILED DESCRIPTION:
Vitamin D is an important nutrient to maintain both skeletal and non-skeletal function. In this study, we have 4 specific aims:

The primary aim of this prospective observational study is to compare the pre- to 6 week, 1 year, 2 year and 5 year post-THA within-patient change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scores between patients who have a low preoperative serum vitamin D level and patients who do not have a low serum vitamin D level. Low serum vitamin D will be defined as serum 25-hydroxy vitamin D level less than 32 ng/ml.

The secondary aim is to compare the pre- to 6 week, 1 year, 2 year and 5 year post-THA within-patient change in performance-based tests (get up and go test, 2 minute walking test) between patients who have a low preoperative serum vitamin D level and patients who do not have a low serum vitamin D level.

The third aim is to compare the pre- to 6 week, 1 year, 2 year and 5 year post-THA within-patient change in Short-form 36 health survey (SF-36) scores between patients who have a low preoperative serum vitamin D level and patients who do not have a low serum vitamin D level.

The fourth aim is to compare the rate of postoperative fracture or thigh pain between patients who have a low preoperative serum vitamin D level and patients who do not have a low serum vitamin D level.

Postoperative thigh pain is defined as pain at the anterolateral aspect of mid thigh which corresponds to the level of the prosthetic stem tip. Thigh pain is characterized by pain in the start-up phase, diminishes during movement and is absent at rest.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 40 and 100 years old, and are scheduled for primary total hip arthroplasty with two surgeons (Drs. Sculco and Cornell) at Hospital for Special Surgery.
* Patients who have a serum 25-OH vitamin D drawn as part of their preoperative work-up.

Exclusion Criteria:

* Bilateral one-stage total hip replacements
* Patients who required a complex surgical procedure including extensive bone grafting, osteotomy, extensive soft tissue release, or a need of adjunctive internal fixation with cables, wires or plate
* Those with serious medical co-morbidities that need adjusted rehabilitation protocol due to their medical problems
* Those who require immediate postoperative revision due to dislocation, infection or component malalignment

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for primary total hip replacement will be identified at the preoperative visit.
Sampling Method: Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2014-02-03 (Actual)

PRIMARY OUTCOMES:
The difference in the within-patient change in WOMAC scores between groups. | preoperatively, 6 week, 1 year, 2 year and 5 year post-THA
  The primary outcome will be the difference in the within-patient change in pre- to 6 week, 1 year, 2 year and 5 year post-THA WOMAC scores between groups. A clinically important difference between groups will be considered as 5 points change in the functional component of WOMAC.
  WOMAC is obtained as part of the HOOS questionnaire which is routinely used in all patients that are scheduled for total joint replacements at Hospital for Special Surgery. We will obtain this score at both pre-operative screening and 6 week, 1 year, 2 year and 5 year after the surgery.

SECONDARY OUTCOMES:
The difference in the within-patient change of the performance-based tests between groups. | preoperatively, 6 weeks, 1 year, 2 years, and 5 years post THA
  Secondary outcome will be the difference in the within-patient change of the performance-based tests (get up and go test and 2 minute walking test) between pre- and 6 week, 1 year, 2 year and 5 year post-THA.
The difference in the within-patient change in SF-36 scores between groups | preoperatively, 6 weeks, 1 year, 2 year, and 5 years postoperatively
  Tertiary outcome will be the difference in the within-patient change in pre- to 6 week, 1 year, 2 year and 5 year post-THA SF-36 scores between groups Preoperative SF-36 is also included as part of the HOOS questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Lane, MD, Principal Investigator — Hospital for Special Surgery, New York; Aasis Unnanuntana, MD, Study Director — Hospital for speicial surgery
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Janssen HC, Samson MM, Verhaar HJ. Vitamin D deficiency, muscle function, and falls in elderly people. Am J Clin Nutr. 2002 Apr;75(4):611-5. doi: 10.1093/ajcn/75.4.611. PMID 11916748
- [Background] Stein MS, Wark JD, Scherer SC, Walton SL, Chick P, Di Carlantonio M, Zajac JD, Flicker L. Falls relate to vitamin D and parathyroid hormone in an Australian nursing home and hostel. J Am Geriatr Soc. 1999 Oct;47(10):1195-201. doi: 10.1111/j.1532-5415.1999.tb05199.x. PMID 10522952
- [Background] Birge SJ. Can falls and hip fracture be prevented in frail older adults? J Am Geriatr Soc. 1999 Oct;47(10):1265-6. doi: 10.1111/j.1532-5415.1999.tb05212.x. No abstract available. PMID 10522964
- [Background] Bischoff HA, Stahelin HB, Urscheler N, Ehrsam R, Vonthein R, Perrig-Chiello P, Tyndall A, Theiler R. Muscle strength in the elderly: its relation to vitamin D metabolites. Arch Phys Med Rehabil. 1999 Jan;80(1):54-8. doi: 10.1016/s0003-9993(99)90307-6. PMID 9915372
- [Background] Mowe M, Haug E, Bohmer T. Low serum calcidiol concentration in older adults with reduced muscular function. J Am Geriatr Soc. 1999 Feb;47(2):220-6. doi: 10.1111/j.1532-5415.1999.tb04581.x. PMID 9988294
- [Background] Bischoff-Ferrari HA, Dietrich T, Orav EJ, Dawson-Hughes B. Positive association between 25-hydroxy vitamin D levels and bone mineral density: a population-based study of younger and older adults. Am J Med. 2004 May 1;116(9):634-9. doi: 10.1016/j.amjmed.2003.12.029. No abstract available. PMID 15093761
- [Background] Gloth FM 3rd, Smith CE, Hollis BW, Tobin JD. Functional improvement with vitamin D replenishment in a cohort of frail, vitamin D-deficient older people. J Am Geriatr Soc. 1995 Nov;43(11):1269-71. doi: 10.1111/j.1532-5415.1995.tb07404.x. PMID 7594162
- [Background] Verhaar HJ, Samson MM, Jansen PA, de Vreede PL, Manten JW, Duursma SA. Muscle strength, functional mobility and vitamin D in older women. Aging (Milano). 2000 Dec;12(6):455-60. doi: 10.1007/BF03339877. PMID 11211956